CLINICAL TRIAL: NCT01685632
Title: Intra Peritoneal Chemo Hyperthermia (IPCH) : Cellular and Metabolic Consequences
Acronym: CHIP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 11-PP-01
Record Dates: First submitted 2012-09-12; First posted 2012-09-14 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Peritoneal Carcinomatosis From Colorectal or Ovarian Origin
Keywords: intra peritonal chemo hyperthermia; peritoneal carcinomatosis; colorectal cancer; ovarian cancer
MeSH Terms: conditions — Peritoneal Neoplasms; Colorectal Neoplasms; Ovarian Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgery with IPCH (Active Comparator): Patients having an IPCH (Intra Peritoneal Chemo Hyperthermia) during the surgery time
  Interventions: Procedure: Surgery with IPCH
- patients without IPCH (Sham Comparator): Patients recused for the surgery due to intraoperative contraindication
  Interventions: Procedure: Without surgery and without IPCH

INTERVENTIONS:
Procedure: Surgery with IPCH — surgical debulking and extensive tumoral resection after laparotomy under general anesthesia
  * 7 blood samples over 72 hours, including 4 samples under general anesthesia throughout surgery and 3 samples during the 3 following days (at 24th, 48th and 72th hours).
  * 6 tissue biopsies, i.e. 2 from peritoneum disease-free and 2 from invaded peritoneum , each representing a volume less than 1 cm3 and 2 biopsies from healthy colonic tissue for the colon-related cancer and 4 biopsies (peritoneum n=2, tumoral tissue n=2) for ovarian-related cancer. All biopsies are done during the surgery under general anesthesia, and each biopsy per site before/after IPCH
  Arms: Surgery with IPCH
Procedure: Without surgery and without IPCH — The patients is opened and recused during the surgery because of extended carcinosis and closed without resection neither IPCH.
  * 7 blood samples over 72 hours, including 4 samples under general anesthesia throughout surgery (2 hours before IPCH, 1.5hours after IPCH, 4 hours after IPCH) and 3 samples during the 3 following days (at 24th, 48th and 72th hours).
  * 6 tissue biopsies, i.e. 2 from peritoneum disease-free and 2 from invaded peritoneum, each representing a volume less than 1 cm3 and 2 biopsies from healthy colonic tissue for the colon-related cancer and 4 biopsies (peritoneum n=2, tumoral tissue n=2) for ovarian-related cancer. All biopsies are done during the surgery under general anesthesia, and each biopsy per site before/after IPCH
  Arms: patients without IPCH

SUMMARY:
Intra Peritoneal Chemo Hyperthermia (IPCH) is a recently validated option for the treatment of peritoneal carcinomatosis from colorectal or ovarian origin. This therapeutic program demonstrated a significant improvement of the late stages (i.e. carcinomatosis) of the disease. From a clinical point of view, within the first 24 hours after IPCH, patients undergo a systemic inflammatory response syndrome, and therefore require to be monitored in an intensive care unit. From a metabolic perspective, preliminary data have been shown a significant "anaerobic style" disturbance of energetic metabolism, suggesting a deep cellular energetic deficit throughout IPCH process.

Putative contradictory effects of IPCH, like the increase of chemotherapy-related cellular toxicity due to heat and on the other hand the initiation of a stress protein response (heat shock response) which helps to reduce the cell injuries, leads to conduct a research project on the underlying mechanisms: consequences, in terms of patient's care and follow-up, are of high relevance.

The primary goal is a multimodal assessment of the IPCH-related cell modifications: signaling pathways, apoptosis and antitumoral immune response.

The assessment criteria include Heat shock protein expression (blood/cell ratio) compared to baseline values, apoptosis and immune response before/after IPCH.

The scheduled sample size is 30 patients having an IPCH and 30 patients contraindicated per surgery.

DETAILED DESCRIPTION:
Intra Peritoneal Chemo Hyperthermia (IPCH) is a recently validated option for the treatment of peritoneal carcinomatosis from colorectal or ovarian origin. This therapeutic program demonstrated a significant improvement of the late stages (i.e. carcinomatosis) of the disease (survival median > 33 months). IPCH induces morbidity as high as 20% and mortality less than 4%. From a clinical point of view, within the first 24 hours after IPCH, patients undergo a systemic inflammatory response syndrome, and therefore require to be monitored in an intensive care unit. From a metabolic perspective, preliminary data have been shown a significant "anaerobic style" disturbance of energetic metabolism, suggesting a deep cellular energetic deficit throughout IPCH process.

Putative contradictory effects of IPCH, like the increase of chemotherapy-related cellular toxicity due to heat and on the other hand the initiation of a stress protein response (heat shock response) which helps to reduce the cell injuries, leads to conduct a research project on the underlying mechanisms: consequences, in terms of patient's care and follow-up, are of high relevance.

Heat shock protein expression (stress protein response markers) and apoptosis are the main chosen tools to evaluate IPCH-related cellular consequences.

Goals of the study Primary goal Multimodal assessment of the IPCH-related cell modifications: signaling pathways, apoptosis and antitumoral immune response.

Secondary goal Comparative study of Heat shock protein expression, whether IPCH is done or the patient is recused for the surgery due to intraoperative contraindication.

Method Prospective cohort follow up Procedure

Besides the usual care (surgical debulking and extensive tumoral resection after laparotomy under general anesthesia), the research protocol includes :

* 7 blood samples over 72 hours (meaning less than 40 ml), including 4 samples under general anesthesia throughout surgery and 3 samples during the 3 following days (at 24th, 48th and 72th hours).
* 6 tissue biopsies, i.e. 2 from peritoneum disease-free and 2 from invaded peritoneum , each representing a volume less than 1 cm3 and 2 biopsies from healthy colonic tissue for the colon-related cancer and 4 biopsies (peritoneum n=2, tumoral tissue n=2) for ovarian-related cancer. All biopsies are done during the surgery under general anesthesia, and each biopsy per site before/after IPCH.

Assessment criteria

* main criteria : Heat shock protein expression (blood/cell ratio) compared to baseline values.
* associate criteria : apoptosis and immune response before/after IPCH Statistical method/Sample size/Study's lenght Scheduled sample size is 30 patients having an IPCH and 30 patients contraindicated per surgery.

The normal distribution is verified using the d'Agostino-Pearson test. For intragroup comparisons, the repeated measures ANOVA is done. For intergroup comparisons, an univariate analysis is done, using the Student t-test and the Fisher exact test.

Taking into account the planned sample size and the annual number of IPCH, the scheduled length of the study is 18 months.

ELIGIBILITY:
Inclusion Criteria:

* adult patient
* eligible for IPCH
* with a social security number
* having a signed an informed consent

Exclusion Criteria:

* study refusal
* parturiants
* psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
heat shock protein expression (blood/cell ratio)compared to baseline values | samples taken under general anesthesia throughout surgery and during the 3 following days (24h, 48h,72h)
  * 7 blood samples over 72 hours (meaning less than 40 ml), including 4 samples under general anesthesia throughout surgery and 3 samples during the 3 following days (at 24th, 48th and 72th hours).
  * 6 tissue biopsies, i.e. 2 from peritoneum disease-free and 2 from invaded peritoneum , each representing a volume less than 1 cm3 and 2 biopsies from healthy colonic tissue for the colon-related cancer and 4 biopsies (peritoneum n=2, tumoral tissue n=2) for ovarian-related cancer. All biopsies are done during the surgery under general anesthesia, and each biopsy per site before/after IPCH.

CONTACTS AND LOCATIONS:
Overall Officials: Michel CARLES, PhD, Principal Investigator — Anesthesia Department, CHU de NICE
Locations (1):
- Département d'Anesthésie Réanimation, CHU de Nice, Nice, France